CLINICAL TRIAL: NCT06773897
Title: The Rutgers University Genetics Coordinating Center Breast Cancer Study
Brief Title: Rutgers University Study of the Genetics of Breast Cancer.
Acronym: RUGCC-BC
Status: Recruiting | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Tara Matise, Ph.D., Distinguished Professor, Rutgers, The State University of New Jersey
Other Study IDs: Pro2023001275
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer Risk; Breast Cancer Prevention; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Health Surveys

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Cancer Cases: Study participants who have been diagnosed with any form of breast cancer, either currently or in the past.
  Interventions: Genetic: Saliva sample; Other: Health Surveys
- Breast Cancer Controls: Study participants who have never had a diagnosis of breast cancer.
  Interventions: Genetic: Saliva sample; Other: Health Surveys

INTERVENTIONS:
Genetic: Saliva sample — Saliva sample is sent via prepaid US Mail for DNA extraction
Other: Health Surveys — Health surveys are filled out online in the study portal.

SUMMARY:
The goal of this observational study is to learn more about how genes impact the risk of breast cancer. Anyone 18 or older living in the US is eligible, and a diagnosis of cancer is NOT required. Study participation is online, and it takes about 20 minutes to complete health surveys and request a saliva collection kit sent through US mail. In return, study participants may opt to receive information about their genetic ancestry at no cost.

DETAILED DESCRIPTION:
This is an online research study to learn more about how genes affect the risk of breast cancer. No office visit is required and in return, participants may receive information about their genetic ancestry for free. BRCA1 and BRCA2 explain only about 25% of the genetic cause of breast cancer. This study will increase our understanding of the genetic basis of breast cancer, which is a crucial step in drug development to improve current treatment options. The study investigators seek a diverse population because men can also get breast cancer and diversity among participants maximizes the usefulness of the data. Participants will use our online study portal to answer questions about their health and provide their DNA via a saliva sample using a pre-paid mailer. Participation takes approximately 20 minutes. Participants will be invited to share data from their electronic health records, but this is not required for study participation. The study investigators keep participants engaged with short monthly newsletters.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* currently living in the United States
* able to understand and follow written instructions in English
* have access to the internet and a computer, laptop, tablet or smart phone
* willing to provide written informed consent for participation
* willing to provide DNA via a saliva sample using a collection kit mailed to the study participant's home
* willing to complete a survey with questions about health related to the study of breast cancer.

Exclusion Criteria:

* Not able to meet or fulfill any of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of anyone at least 18 years old who lives in the United States, including both individuals who have or had breast cancer and those who have not. Participants include males, females, non-binary, and all race-ethnic groups.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Genetic risk variants associated with breast cancer | 2 years
  Genetic factors will be measured through whole exome sequencing along with genotyping of common variants, and then correlated with breast cancer and breast cancer subtype.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Matise, Ph.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers University, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study website with detailed information about the study. — https://rugcc.rutgers.edu/breast_cancer/
- See also: Study portal for participant enrollment and study engagement. — https://go.rutgers.edu/BCStudyCTG